CLINICAL TRIAL: NCT04932096
Title: Sleep Management And Recovery After Traumatic Brain Injury in Kids (SMARTKids): Evidence for Targeting Sleep to Improve Outcomes
Brief Title: Sleep Management And Recovery After Traumatic Brain Injury in Kids: Pilot Intervention of Melatonin
Acronym: SMARTKids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cydni Williams, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPEDI1282A; 1K23HL150229-01A1 (NIH)
Record Dates: First submitted 2021-06-02; First posted 2021-06-18 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury; Critical Illness; Sleep
Keywords: pediatric; traumatic brain injury; melatonin; sleep; intervention
MeSH Terms: conditions — Brain Injuries, Traumatic; Critical Illness | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): (melatonin doses of 3mg or 5mg based on patient size given nightly 1 hour prior to bedtime every night for 30 days)
  Interventions: Drug: melatonin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: melatonin — melatonin supplementation
  Arms: Melatonin
Other: placebo — microcrystalline cellulose filled capsule
  Arms: Placebo

SUMMARY:
Sleep wake disturbances compound recovery in over half of pediatric traumatic brain injury survivors, leading to impaired quality of life, and few effective interventions exist to treat this important morbidity. Therefore, this study will conduct a randomized controlled trial evaluating a melatonin intervention started during hospitalization and continued after discharge compared to placebo. The trial will investigate if this intervention is feasible, acceptable, and effective at reducing sleep wake disturbances as measured on the Sleep Disturbances Scale for Children 1-month after hospital discharge.

Participants will be randomly assigned to receive the intervention (melatonin) or to the control group (placebo) with a goal of equal numbers of participants in each group and all will receive sleep education. Participants will be followed closely after consent and outcomes will be assessed at hospital discharge, and 1-month. Outcomes will focus on feasibility (ability to recruit patients into the trial) and acceptability (patient safety and satisfaction), but will also assess the effectiveness of the intervention to reduce sleep disturbances after discharge. The investigators will assess sleep using questionnaires and actigraphy (watch-like activity monitors). Exploratory outcomes will include global health outcomes.

ELIGIBILITY:
Inclusion:

* Children age ≥6 years and <19 years
* Traumatic brain injury defined as disruption of the normal function of the brain resulting from blunt force injury with a severity defined as mild complicated, moderate, or severe by the Glasgow Coma Scale with the presence of intracranial injury on imaging
* Admission to Oregon Health & Science University Hospitals
* Deemed likely to survive hospitalization by clinical care team
* Able to tolerate enteral medications within 72 hours of admission
* Child participant resides with parent or legal guardian

Exclusion:

* Lack stable means of communication with study team (phone, email, mailing address)
* Abusive trauma suspected or confirmed
* Dialysis
* Extracorporeal support (e.g. ECMO)
* Significant liver injury defined as >2x normal levels for AST or ALT
* Clinical team safety concerns with use of intervention
* Pregnancy
* Prisoners

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cydni Williams, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Basic tabular results will be entered into clinicaltrials.gov within 1 year of primary completion of the study. We will make participant data available to researchers once thoroughly de-identified and approved by our institutional review board within 1 year of study completion. Data will be made available on requests made directly to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol and SAP will be shared upon approval by the Institutional Review Board, and the final approved study protocol and SAP with documentation of any amendments will be available at study completion. The ICF will be shared no later than 60days from enrollment of the last study visit. A CSR and analytic code for the primary outcomes analysis will be made available within 1 year of study completion.
Access Criteria: Requests for data can be made by contacting the Principal Investigator

REFERENCES:
- [Background] Luther M, Poppert Cordts KM, Williams CN. Sleep disturbances after pediatric traumatic brain injury: a systematic review of prevalence, risk factors, and association with recovery. Sleep. 2020 Oct 13;43(10):zsaa083. doi: 10.1093/sleep/zsaa083. PMID 32328648
- [Background] Poppert Cordts KM, Hall TA, Hartman ME, Luther M, Wagner A, Piantino J, Guilliams KP, Guerriero RM, Jara J, Williams CN. Sleep Measure Validation in a Pediatric Neurocritical Care Acquired Brain Injury Population. Neurocrit Care. 2020 Aug;33(1):196-206. doi: 10.1007/s12028-019-00883-5. PMID 31797275
- [Background] Williams CN, Hartman ME, McEvoy CT, Hall TA, Lim MM, Shea SA, Luther M, Guilliams KP, Guerriero RM, Bosworth CC, Piantino JA. Sleep-Wake Disturbances After Acquired Brain Injury in Children Surviving Critical Care. Pediatr Neurol. 2020 Feb;103:43-51. doi: 10.1016/j.pediatrneurol.2019.08.010. Epub 2019 Aug 26. PMID 31735567
- See also: Principal Investigator program website that will be updated regularly for PI contact information and study related materials — http://www.ohsu.edu/pccnrp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 of 53 eligible and approached participants recruited between January 2, 2023 and March 1, 2025. All participants were recruited during hospitalization for traumatic brain injury.
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 10 | 11
Completed | 9 | 9
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Partial completion (did not complete primary outcome survey) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10.3 [9.7 to 13.6] | 12.8 [7.7 to 14.8] | 10.7 [8.3 to 14.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 1 | 3
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Medicaid Insurance Status [Count of Participants; unit: Participants]
  Medicaid | 6 | 6 | 12
  Private Insurance | 4 | 5 | 9
Admission Glasgow Coma Scale Score [Count of Participants; unit: Participants]
  Mild, score 13-15 | 7 | 9 | 16
  Moderate, score 9-12 | 1 | 0 | 1
  Severe, score 3-8 | 2 | 2 | 4
Pre-injury medical condition present [Count of Participants; unit: Participants] | 3 | 2 | 5
Pre-injury psychological diagnosis present [Count of Participants; unit: Participants] | 0 | 1 | 1
Pre-injury neurodevelopmental condition present [Count of Participants; unit: Participants] | 3 | 3 | 6
Skull fracture present at admission [Count of Participants; unit: Participants] | 9 | 6 | 15
Intracranial injury on imaging present at admission [Count of Participants; unit: Participants] | 8 | 6 | 14
Other injuries (non-brain) present at admission [Count of Participants; unit: Participants] | 3 | 6 | 9
Inpatient Rehabilitation Discharge Disposition [Count of Participants; unit: Participants] | 1 | 0 | 1
Sleep Disturbances Scale for Children Total score [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5 for a range of possible total scores of 26 - 130. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction, and T-scores greater than 60 generally indicating clinically significant dysfunction.
  T-score | 60 [55 to 64] | 63 [56 to 76] | 60 [48.5 to 74.5]
Sleep Disturbances Scale for Children Initiation and Maintenance Subscale [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction. T-scores greater than 60 generally indicating clinically significant dysfunction. The Disorders of Initiation and Maintenance Subscale evaluates potential disorders like insomnia or circadian rhythm disturbances.
  T-score | 64 [47 to 76] | 76 [64 to 79] | 66 [52 to 79]
Sleep Disturbances Scale for Children Breathing Subscale [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction. T-scores greater than 60 generally indicating clinically significant dysfunction. The Breathing Subscale evaluates potential disorders like sleep apnea.
  T-score | 51 [45 to 64] | 51 [51 to 58] | 51 [45 to 61]
Sleep Disturbances Scale for Children Arousal Subscale [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction. T-scores greater than 60 generally indicating clinically significant dysfunction. The Arousal subscale evaluates potential disorders like sleepwalking and night terrors.
  T-score | 47 [47 to 47] | 47 [47 to 58] | 47 [47 to 58]
Sleep Disturbances Scale for Children Sleep Wake Transition Subscale [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction. T-scores greater than 60 generally indicating clinically significant dysfunction. The sleep wake transition subscale evaluates potential disorders like sleep talking or sleep movement disorders.
  T-score | 62 [50 to 66] | 50 [50 to 70] | 54 [45 to 68]
Sleep Disturbances Scale for Children Somnolence Subscale [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction. T-scores greater than 60 generally indicating clinically significant dysfunction. The somnolence subscale evaluates potential disorders of excessive sleepiness or narcolepsy.
  T-score | 50 [46 to 53] | 50 [50 to 64] | 50 [44 to 66.5]
Sleep Disturbances Scale for Children Hyperhidrosis Subscale [Median (Inter-Quartile Range); unit: T-score] — Sleep Disturbances Scale for Children: 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5. Raw scores are converted to measured defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating dysfunction. T-scores greater than 60 generally indicating clinically significant dysfunction. The hyperhidrosis subscale evaluates excessive sweating during sleep.
  T-score | 45 [45 to 45] | 45 [45 to 58] | 45 [45 to 54.5]

OUTCOME MEASURES:

1. Primary Outcome: Sleep Disturbances Scale for Children
Description: Sleep Disturbances Scale for Children (SDSC): 26-item parent proxy sleep questionnaire with higher scores reflecting greater disturbance and risk for clinically important sleep disorders. Each question is scored 1 through 5 for a range of possible total scores of 26 - 130. Raw scores are converted to measure defined T-scores (mean=50, SD=10) for the total score and 6 subscale scores with higher scores indicating worse dysfunction, and T-scores greater than 60 generally indicating clinically significant dysfunction in the total score and all 6 subscale scores. The subscales include Initiation and Maintenance, Arousal, Breathing, Transition, Somnolence, and Hyperhidrosis.
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
T-score
  Total T-score | 55 [47 to 68] | 69 [63 to 79]
  Initiation and Maintenance T-score | 64 [50 to 89] | 73 [64 to 79]
  Breathing T-score | 51 [45 to 51] | 58 [51 to 58]
  Arousal T-score | 47 [47 to 47] | 58 [47 to 58]
  Transition T-score | 50 [50 to 54] | 54 [50 to 79]
  Somnolence T-score | 50 [50 to 50] | 62 [53 to 73]
  Hyperhidrosis T-Score | 45 [45 to 51] | 45 [45 to 45]

2. Primary Outcome: Recruitment
Description: Quantitative number of patients consented per patients approached
Time Frame: through study completion, an average of 6-months
Population: Number of eligible patients approached for consent
Measure: Count of Participants; unit: Participants
Groups:
- Approached Patients: All hospitalized trauma patients meeting inclusion/exclusion criteria approached for consent
Arm/Group | Approached Patients
Number analyzed (Participants) | 53
Participants | 21

3. Primary Outcome: Retention
Description: Quantitative number of participants completing trial procedures per patients consented
Time Frame: through study completion, an average of 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Completion of Study Procedures: Number of patients completing study procedures
Arm/Group | Completion of Study Procedures
Number analyzed (Participants) | 21
Participants
  Completion of Sleep Disturbances Scale for Children Survey | 18
  Completion of other procedures but not Sleep Disturbances Scale for Children survey | 1
  Participant withdrawal from study | 2

4. Secondary Outcome: Adherence Quantitative
Description: pill counts, report of using study medication at least 5/7 days per week
Time Frame: 1-month
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
Participants | 8 | 7

5. Secondary Outcome: Adherence Qualitative
Description: participant report of compliance with treatment regimen evaluated by survey question estimating percentage of study days compliant with intervention
Time Frame: 1-month
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
Participants | 8 | 7

6. Secondary Outcome: Pediatric Quality of Life Inventory Multidimensional Fatigue Scale
Description: Pediatric Quality of Life Inventory Multidimensional Fatigue Scale (PedsQL MFS); 18 item parent proxy report of fatigue using a likert scale. Responses to each question receive a score of 0, 25,50,75, or 100. The measure provides a total score and three subscale scores- General, Sleep/rest, and Cognitive fatigue subscales based on the average response to each question for the total score and the average response to each subscale's questions for the subscale scores. All scores (total and subscale) range 0-100 with higher scores indicating better function and less fatigue.
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale
  Total Score | 63.9 [58.3 to 83.3] | 54.9 [43.8 to 76.4]
  General Fatigue Subscale | 70.8 [62.5 to 79.2] | 50 [37.5 to 87.5]
  Sleep/rest Fatigue Subscale | 70.8 [50 to 83.3] | 58.3 [33.3 to 85.4]
  Cognitive Fatigue Subscale | 75 [63 to 79.2] | 54.1 [47.9 to 77.1]

7. Secondary Outcome: Chronotype
Description: Children's Chronotype Questionnaire, parent reported survey of circadian rhythm characteristics. Morningness/Eveningness Scale Score summed from responses, range 10 (morningness) to 49 (eveningness)
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 24.5 [22 to 26.5] | 25 [21 to 28]

8. Secondary Outcome: Sleep Latency
Description: actigraphy measured time in minutes to fall asleep
Time Frame: 1-month
Population: Actigraphy usable providing 5/7 days per week of data
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
minutes | 4.6 [3.9 to 7.2] | 5.3 [2.7 to 12.4]

9. Secondary Outcome: Total Sleep Time
Description: actigraphy measured total time asleep in minutes
Time Frame: 1-month
Population: Actigraphy usable data if 5/7 days per week
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
minutes | 471 [446 to 475] | 459 [413 to 496]

10. Secondary Outcome: Wake After Sleep Onset
Description: actigraphy measured time in minutes awake after sleep onset
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
minutes | 4.4 [4.2 to 4.5] | 4.2 [3 to 4.9]

11. Secondary Outcome: Number of Night Awakenings
Description: actigraphy measured number of instances awoken after sleep onset
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: number of awakenings
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
number of awakenings | 31.2 [28.9 to 34.5] | 30.5 [26.9 to 32.4]

12. Secondary Outcome: Sleep Efficiency
Description: actigraphy measure percentage of nighttime period spent asleep
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: percentage of time in bed deemed asleep
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
percentage of time in bed deemed asleep | 88 [87.3 to 88.1] | 88 [87.2 to 88.4]

13. Secondary Outcome: Sleep Onset Time
Description: time of day fell asleep presented as hours corresponding the the time of day from midnight as 0 hours (e.g., 22.5 hours means they fell asleep at 10:30 pm)
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: hours corresponding to time of day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
hours corresponding to time of day | 23.42 [23.13 to 23.42] | 22.77 [22.28 to 23.78]

14. Secondary Outcome: Sleep Offset Time
Description: time of day waking from nighttime sleep presented in hours from midnight as time 0 (e.g., 7.5 hours means they woke up at 7:30 am)
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: hours corresponding to time of day
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
hours corresponding to time of day | 8.28 [7.97 to 8.52] | 7.58 [6.45 to 7.83]

15. Secondary Outcome: Adverse Events Time 0
Description: Evaluation of adverse events asking participants to report any side effects of study interventions; Number of patients with any adverse event reported or noted on symptom screening checklist
Time Frame: hospital discharge assessed up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 10 | 11
Participants
  Readmission to hospital, not study related | 1 | 0
  EVD placement and hyponatremia, not study related | 1 | 0
  Nausea, vomiting at discharge | 0 | 1
  headaches at discharge | 0 | 1
  None | 8 | 9

16. Secondary Outcome: Adverse Events Time 1
Description: Evaluation of adverse events asking participants to report any side effects of study interventions
Time Frame: 1-month
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Reason for Non-adherence
Description: qualitative response to survey question about reasons for non-compliance with treatment regimen or sleep plan
Time Frame: 1-month
Population: Reasons given for not using study medication every night or sleep plan resources at any frequency
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 7 | 8
Participants
  Misplaced medication | 1 | 0
  Pharmacy issues | 0 | 1
  Patient wanted to stop medication | 0 | 1
  Transitioning between parent houses or moving | 1 | 1
  Fell asleep before taking medication | 1 | 1
  forgot about sleep education | 2 | 2
  Did not see sleep education in paperwork | 2 | 2

18. Other Pre Specified Outcome: Health Related Quality of Life
Description: Pediatric Quality of Life Inventory (PedsQL): parent reported measure of quality of life. Scores range 0-100 with higher scores indicating better quality of life.
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 71.7 [63 to 73.2] | 59.8 [48.9 to 79.9]

19. Other Pre Specified Outcome: Cognitive Functioning
Description: Behavior Rating Inventory of Executive Function, second edition (BRIEF-2); parent proxy report of everyday executive function, reported as standardized Global Executive Composite T-score, with higher scores indicating worse function. T-scores range from 0-100, with a mean of 50 and standard deviation of 10.
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: T-score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
T-score on a scale | 52 [45 to 59] | 55 [46 to 60]

20. Other Pre Specified Outcome: Physical Functioning
Description: Functional Status Scale, range 6-30, with higher scores indicating worse function; measured at followup
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 6 [6 to 6] | 6 [6 to 6]

21. Other Pre Specified Outcome: Anxiety
Description: Patient Reported Outcome Measurement Information System (PROMIS) anxiety short form T-score with higher scores indicating worse outcome. T-scores range from 0 - 100, with a mean of 50 and standard deviation of 10.
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: T-score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
T-score on a scale | 38 [34 to 45] | 50 [41 to 55]

22. Other Pre Specified Outcome: Depression
Description: Patient Reported Outcome Measurement Information System (PROMIS) depression short form T-score with higher scores indicating worse outcome. T-scores range from 0-100, with a mean of 50 and standard deviation of 10.
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: T-score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
T-score on a scale | 45 [36 to 57] | 47 [39 to 51]

23. Other Pre Specified Outcome: PROMIS Pain Behavior
Description: Patient Reported Outcome Measurement Information System (PROMIS) pain behavior (T-score with mean of 50 and standard deviation of 10) parent report forms; Higher scores indicate worse pain outcomes
Time Frame: 1-month
Measure: Median (Inter-Quartile Range); unit: T-score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 9 | 9
T-score on a scale | 47 [42 to 51] | 10 [10 to 36]

ADVERSE EVENTS:
Time Frame: 30 days and up to 47 days after study start to complete survey
Description: Symptom checklist assessed at follow up visit.
Groups:
- Melatonin: melatonin doses of 3mg or 5mg based on patient size given nightly 1 hour prior to bedtime every night for 30 days; this arm is not separated by dose administered as all patients received weight based dosing per standard practice in pediatrics
  melatonin: melatonin supplementation
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin (N=10) | Placebo (N=11)
Readmission to hospital (Nervous system disorders) | 1 (1) | 0 (0) — Patient readmitted to hospital for injury related complications, deemed not related to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin (N=10) | Placebo (N=11)
Fatigue (General disorders) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 2 (2) | 2 (2)
Behavior change with increased anxiety (General disorders) | 0 (0) | 2 (2)
double vision (Eye disorders) | 1 (1) | 0 (0)
motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
nightmares (Psychiatric disorders) | 1 (1) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Appetite change (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot trial with small number of participants recruited. Results focus on feasibility, was not powered to detect differences in sleep and other secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04932096/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04932096/ICF_001.pdf